CLINICAL TRIAL: NCT05895292
Title: Digital Analysis of Denture Space Confines and Patient's Satisfaction for Conventional Versus Neutral-Zone CAD/CAM Dentures Restoring Mandibular Resorbed Ridges.(Randomized Controlled Clinical Trial)
Brief Title: Conventional Versus Neutral-Zone CAD/CAM Dentures Restoring Mandibular Resorbed Ridges
Acronym: CAD/CAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnia M. Refai, Lecturer of Oral and Maxillofacial Prosthodontics,faculty of dentistry , Ain Shams university, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecIR012316
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Denture, Complete
Keywords: CAD/CAM; Denture, Complete; Patient Satisfaction; Dental Impression Technique
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Twelve patients will be randomly assigned to one of two groups (I or II) by a practitioner who will not be involved in patient selection or treatment but will be aware of the randomization sequence and have access to the randomization lists. This will be stored on a password-protected laptop, and the randomly generated codes will be placed in sequentially ordered, opaque, and sealed envelopes using a research randomizer (https://www.randomizer.org/). Participants were randomized to first receiving either Conventional CAD/CAM manufactured complete removable dentures Based on bone support concept or CAD/CAM neutral zone complete dentures will be designed based on the neutral zone concept and then after 3 months cross over to the other set. Patients and clinical practitioners are blinded to the type of prostheses at all study times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM Milled Methacrylate Complete Removable Dentures based on bone-support concept. (Experimental): The patient will be provided by a complete removable denture designed according to bone-support concept to restore his missing teeth which will be manufactured by CAD/CAM milling of monolithic methacrylate blanks.
  Interventions: Device: CAD/CAM Milled Methacrylate Complete Removable Dentures based on bone-support concept.
- CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept. (Active Comparator): The patient will be provided with a complete removable denture designed according to the neutral-concept to restore his missing teeth, which will be manufactured by CAD/CAM milling of monolithic methacrylate blanks.
  Interventions: Device: CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept.

INTERVENTIONS:
Device: CAD/CAM Milled Methacrylate Complete Removable Dentures based on bone-support concept. — The patients will receive complete removable dentures designed based on the bone-support concept and digitally manufactured using a milling machine.
  Arms: CAD/CAM Milled Methacrylate Complete Removable Dentures based on bone-support concept.
Device: CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept. — The patients will receive complete removable dentures designed based on the neutral-zone concept and digitally manufactured using a milling machine
  Arms: CAD/CAM Milled Methacrylate Complete Removable Dentures based on neutral zone concept.

SUMMARY:
The study is a within-subject randomized clinical trial that will compare and evaluate patients' satisfaction and digitally analyze denture space Confines. Group I: CAD/CAM. (computer-aided design/computer-aided manufacturing) Conventional complete dentures will be designed based on the bone support concept, Group II: CAD/CAM neutral zone complete dentures will be designed based on the neutral zone concept. The participants will be selected according to inclusion and exclusion criteria and will be randomly allocated into both groups and then shuffled to the other group using the Research Randomizer Program.

DETAILED DESCRIPTION:
This study is designed as a randomized clinical trial applying a within-subject comparison of two different complete denture types as follows; group I: CAD/CAM conventional complete dentures will be designed based on the bone support concept, group II: CAD/CAM neutral zone complete dentures will be designed based on the neutral zone concept. The study will be carried out on twelve completely edentulous patients exhibiting advanced residual ridge resorption, each patient will receive two sets of complete dentures in a random sequence, and each set of CDs will be worn for at least eight weeks after the last recall visit before assessments. Upon delivery of the second set of CDs, the first set will be withheld from the patient. For each denture set, patient satisfaction will be rated using a patient denture assessment PDA questionnaire that will be assessed via a Likert scale, the obtained scores will be used to compare the two denture types. Also by using special digital software, a comparison between group I and II virtual complete denture images will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been completely edentulous in both jaws (maxilla and mandible) for a long period.
2. The age of patients ranges from 50 to 80 years old.
3. Patients with a resorbed mandibular ridge.
4. Patients with a Class I maxillo-mandibular relationship
5. Patients with adequate inter-arch space.
6. Patients with good neuromuscular control.
7. Patients without any tempo-mandibular disorder.

Exclusion Criteria:

1. Patients with any oral diseases that may affect complete denture construction
2. Patients with bad oral hygiene.
3. Patients with oral parafunctional habits.
4. Hysterical patients.
5. Patients will undergo or have previously received chemotherapy or radiotherapy.
6. Drug-addicted patients.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Digital Analysis and Comparison of Denture Space Confines for CAD/CAM Dentures Based on the bone-support concept Versus based on the neutral-zone concept Restoring Mandibular Resorbed Ridges using "Medit compare" digital software. | before manufacturing of complete removable denture
  comparing the position of the neutral zone to the software-designed anatomical denture confines using "Medit compare" digital software (Medit design, Medit Compare (V1.2), Seoul, South Korea). Average values of facio-lingual deviations between the two dentures in the premolar and molar regions, as well as the anterior region, will be calculated in millimeters, yielding five measurements for each patient's denture sets. Color maps for dimensional deviations of the overall as well as specified surfaces for both dentures revealing the qualitative 3D differences between them will be obtained. Measuring procedures will be similar, as recommended by the manufacturer and all will be performed by the same digital professional operator.

SECONDARY OUTCOMES:
Evaluation of patients' satisfaction with both types of the Complete Removable Dentures | three months
  Evaluation of patients' satisfaction with both types of the Complete Removable Dentures by using Patient's Denture Assessment questionnaire (PDA) and interpreting it by using Likert scale (higher score (scale no.5) indicates good outcome and lower score (scale no.1)indicates bad outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain shams University, Cairo, Nasr City, Egypt

REFERENCES:
- [Background] Bhorgonde D, Nandakumar K, Khurana PR, Kumari VS, Reddy MS, Siddique S. An evaluation of the position of the neutral zone in relation to the crest of mandibular alveolar ridge - An In-vivo study. J Int Oral Health. 2014 Apr;6(2):45-54. Epub 2014 Apr 26. PMID 24876702
- [Background] Choi S, Kim S, Chang JS. The Neutral Zone Approach with CAD-CAM Record Bases. J Prosthodont. 2022 Jul;31(6):459-463. doi: 10.1111/jopr.13502. Epub 2022 Mar 24. PMID 35271758